CLINICAL TRIAL: NCT02459665
Title: Preparing for a Clinical Trial of Interventions to Maintain Normal Vaginal Microbiota for Preventing Adverse Reproductive Health Outcomes in Africa
Brief Title: Rwanda Vaginal Microbiota Restoration Study
Acronym: VMB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Janneke van de Wijgert (Other)
Collaborators: Rinda Ubuzima, Rwanda (Unknown)
Responsible Party: Sponsor-Investigator, Janneke van de Wijgert, Professor of Infection and Global Health, University of Liverpool
Organization: University of Liverpool (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: RETH000828
Record Dates: First submitted 2015-05-21; First posted 2015-06-02 (Estimated); Results first posted 2019-07-16 (Actual); Last update posted 2019-07-16 (Actual); Status verified 2019-06

CONDITIONS: Bacterial Vaginosis
MeSH Terms: conditions — Vaginosis, Bacterial

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Group 1 (No Intervention): Negative control group: After initial treatment for BV/TV, no intervention.
- Group 2 (Other): Positive control group: After initial treatment for BV/TV, metronidazole pills (500 mg) twice per week for 2 months.
  Interventions: Drug: Prophylactic use of metronidazole pills (500 mg)
- Group 3 (Active Comparator): After initial treatment for BV/TV, Ecologic Femi+ vaginal capsule (a vaginal probiotic) once per day for 5 days immediately after the initial treatment followed by thrice weekly for two months.
  Interventions: Biological: Vaginal multiple lactobacilli-containing probiotic for prevention of BV recurrence
- Group 4 (Active Comparator): After initial treatment for BV/TV, Gynophilus LP vaginal tablet (a vaginal probiotic) once every 4 days for two months.
  Interventions: Biological: Vaginal Lcr35-containing probiotic for prevention of BV recurrence

INTERVENTIONS:
Biological: Vaginal multiple lactobacilli-containing probiotic for prevention of BV recurrence — Vaginal probiotic to restore the vaginal microbiome and prevent BV recurrence after metronidazole treatment for BV or TV
  Other Names: Ecologic Femi+ vaginal capsule
  Arms: Group 3
Drug: Prophylactic use of metronidazole pills (500 mg) — Prophylactic use of metronidazole pills to prevent BV recurrence after metronidazole treatment for BV or TV
  Other Names: Tricozole
  Arms: Group 2
Biological: Vaginal Lcr35-containing probiotic for prevention of BV recurrence — Vaginal probiotic to restore the vaginal microbiome and prevent BV recurrence after metronidazole treatment for BV or TV
  Other Names: Gynophilus LP vaginal tablet
  Arms: Group 4

SUMMARY:
A pilot randomized controlled clinical trial of intermittent use of two different vaginal lactobacilli-containing probiotics, and oral metronidazole, to prevent bacterial vaginosis recurrence.

DETAILED DESCRIPTION:
This is a pilot study to prepare for larger clinical trials. Sixty-eight HIV-negative, non-pregnant, sexually active women aged 18-45 with bacterial vaginosis (BV, by modified Amsel criteria and/or Nugent score) and/or Trichomonas vaginalis (TV, on wet mount or by culture) will be treated using oral metronidazole for 7 days. After successful treatment, and when they are free of vaginal candidiasis, other curable sexually transmitted infections (STIs) and urinary tract infection (UTI)), they will be randomised to 4 different vaginal microbiome (VMB) maintenance interventions (17 per group) within 3 days of completing oral metronidazole treatment: 1) Behavioral 'vaginal practices cessation and safer sex' counselling only (control); 2) Behavioral counselling plus 500mg metronidazole pills twice per week for two months; 3) Behavioral counselling plus Ecologic Femi vaginal capsule, once per day for 5 days immediately after oral metronidazole treatment followed by thrice weekly, for two months; 4) Group 4: Behavioral counselling plus Gynophilus vaginal tablet, once every 4 days for two months. Vaginal probiotic use may be ceased temporarily during menstruation. Participants will be asked to adhere to the interventions for 2 months, and VMB assessments will take place before (screening and enrolment visits), during (Day 7, Month 1 and Month 2 visits), and after the interventions (Month 6 visit).

ELIGIBILITY:
Inclusion Criteria:

* Sexually active, defined as having had sex at least twice in the two weeks prior to screening
* At high risk of HIV/STIs/BV, defined as having had more than one sexual partner in the last 12 months OR having been treated for an STI and/or BV in the last 12 months
* Successfully treated for BV (modified Amsel criteria) or TV (wet mount), and free of STIs, symptomatic vaginal candidiasis and UTI at enrollment
* Currently in good physical and mental health as judged by a study physician
* Willing and able to adhere to study procedures and provide written informed consent.

Exclusion Criteria:

* Pregnant
* HIV positive
* Clinician-observed genital ulcers, condylomata, or other genital abnormalities at screening or enrollment
* Underwent a gynaecological surgery/invasive procedure in the 3 months prior to screening
* History of significant urogenital prolapse, undiagnosed vaginal bleeding, urine or faecal incontinence, or blood clotting disorders
* Allergic to metronidazole or any other components of the study drugs
* Not willing to stop use of other oral or vaginal probiotics from the screening visit until the end of study participation
* Participating in another health intervention study
* For any other reason potentially interfering with participant safety or protocol adherence as judged by the Principal Investigator

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 68 (Actual)
Dates: Start 2015-06-05 (Actual); Primary Completion 2016-02-23 (Actual); Study Completion 2018-08-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janneke H van de Wijgert, PhD, Study Chair — University of Liverpool

REFERENCES:
- [Derived] Verwijs MC, Agaba S, Umulisa MM, van de Wijgert JHHM. Feasibility and acceptability of frequent vaginal self-sampling at home by Rwandan women at high risk of urogenital tract infections. Sex Transm Infect. 2022 Feb;98(1):58-61. doi: 10.1136/sextrans-2020-054816. Epub 2021 Jan 29. PMID 33514681
- [Derived] Verwijs MC, Agaba S, Umulisa MM, Uwineza M, Nivoliez A, Lievens E, van de Wijgert JHHM. Vaginal probiotic adherence and acceptability in Rwandan women with high sexual risk participating in a pilot randomised controlled trial: a mixed-methods approach. BMJ Open. 2020 May 19;10(5):e031819. doi: 10.1136/bmjopen-2019-031819. PMID 32434932
- [Derived] Verwijs MC, Agaba SK, Darby AC, van de Wijgert JHHM. Impact of oral metronidazole treatment on the vaginal microbiota and correlates of treatment failure. Am J Obstet Gynecol. 2020 Feb;222(2):157.e1-157.e13. doi: 10.1016/j.ajog.2019.08.008. Epub 2019 Aug 9. PMID 31404542

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The target population was women at high risk of urogenital infections living in Kigali, Rwanda. Recruitment activities were implemented by study staff with the help of Community Mobilizers, who were selected due to their strong connections with high-risk women in Kigali. They helped staff organize recruitment meetings in relevant communities.
Pre-assignment Details: At the end of the screening process, women were either ineligible or diagnosed with bacterial vaginosis (by modified Amsel criteria and/or Nugent score) and/or trichomoniasis (by culture or wet mount) and treated with 500 mg oral metronidazole 2x/day for 7 days. An enrollment visit was scheduled within three days after treatment completion.
Groups:
- Control: Behavioral counseling only
- Oral Metronidazole: Oral metronidazole 2-month intermittent use plus counseling
- Ecologic Femi+: Ecologic Femi+ vaginal probiotic capsule 2-month intermittent use plus counseling
- Gynophilus LP: Gynophilus LP vaginal probiotic tablet 2-month intermittent use plus counseling
Period: Overall Study
Arm/Group | Control | Oral Metronidazole | Ecologic Femi+ | Gynophilus LP
Started (Enrollment visit) | 17 | 17 | 17 | 17
Day 7 Visit | 17 | 17 | 17 | 16
Month 1 Visit | 17 | 17 | 17 | 16
Month 2 Visit (Cessation of interventions) | 17 | 16 | 17 | 16
Month 6 Visit (Final study visit) | 17 | 16 | 16 | 15
Completed (Month 6) | 17 | 16 | 16 | 15
Not Completed | 0 | 1 | 1 | 2
Not completed — Withdrawal by Subject | 0 | 1 | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control | Oral Metronidazole | Ecologic Femi+ | Gynophilus LP | Total
Number analyzed (Participants) | 17 | 17 | 17 | 17 | 68
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 17 | 17 | 17 | 17 | 68
  >=65 years | 0 | 0 | 0 | 0 | 0
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 29 [24 to 36] | 30 [27 to 34] | 33 [28 to 35] | 31 [27 to 35] | 31 [27 to 35]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 17 | 17 | 17 | 68
  Male | 0 | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  African (Rwandan) | 17 | 17 | 17 | 17 | 68
Region of Enrollment [Count of Participants; unit: Participants]
  Rwanda | 17 | 17 | 17 | 17 | 68
Exchanged sex for money/goods in past month [Count of Participants; unit: Participants] | 17 | 14 | 15 | 17 | 63
Sex partners in the past month [Median (Inter-Quartile Range); unit: sex partners] | 5 [3 to 20] | 5 [2 to 10] | 3 [2 to 15] | 3 [2 to 20] | 5 [2 to 18]

OUTCOME MEASURES:

1. Primary Outcome: Bacterial Vaginosis (BV) Incidence by Modified Amsel Criteria
Description: Modified Amsel criteria positive is at least 2 of 3 of the following positive: clue cells, vaginal pH, whiff test.
  Modified intent-to-treat (ITT) analyses (women with Nugent 7-10 at enrollment excluded), using person-years (PY) at risk as denominator of each incidence rate.
Time Frame: 2 months (intervention period)
Population: Modified ITT population: all randomized women except women with Nugent 7-10 at enrollment.
Measure: Number (95% Confidence Interval); unit: Incidence: events per PY at risk
Groups:
- Oral Metronidazole: Oral metronidazole 2-months intermittent use plus counseling
- Ecologic Femi+: Ecologic Femi+ vaginal probiotic capsules 2-months intermittent use plus counseling
- Gynophilus LP: Gynophilus LP vaginal probiotic tablets 2-months intermittent use plus counseling
Arm/Group | Control | Oral Metronidazole | Ecologic Femi+ | Gynophilus LP
Number analyzed (Participants) | 15 | 11 | 14 | 11
Incidence: events per PY at risk | 7.53 [4.28 to 13.26] | 2.04 [0.66 to 6.31] | 3.36 [1.51 to 7.48] | 3.35 [1.26 to 8.92]

2. Primary Outcome: Bacterial Vaginosis (BV) Incidence by Nugent Scoring (Nugent 7-10)
Description: The Nugent score is a scale from 0-10 based on visualisation of three different bacterial morphotypes on a Gram stained slide, but in the incidence rates, the variable was used as a binary variable: BV present (Nugent score 7-10) or absent (Nugent score 0-6). Modified intent-to-treat (ITT) analyses (women with Nugent 7-10 at enrollment excluded), using person-years (PY) at risk as the denominator for each incidence rate.
Time Frame: 2 months (intervention period)
Population: Modified ITT population: All randomized women except women with Nugent 7-10 at enrollment.
Measure: Number (95% Confidence Interval); unit: Incidence: events per PY at risk
Arm/Group | Control | Oral Metronidazole | Ecologic Femi+ | Gynophilus LP
Number analyzed (Participants) | 15 | 11 | 14 | 11
Incidence: events per PY at risk | 10.18 [5.48 to 18.92] | 1.41 [0.35 to 5.62] | 3.58 [1.61 to 7.96] | 5.36 [2.41 to 11.93]

3. Primary Outcome: Trichomonas Vaginalis (TV) Incidence by Culture
Description: A swab was inoculated into an InPouch culture pouch, specifically designed for TV growth. The pouch was checked daily for five days to detect growth. The results was positive when growth detected and negative when no growth detected on the fifth day.
  Intent-to-treat (ITT) analyses, using person-years (PY) at risk as the denominator for each incidence rate.
Time Frame: 2 months (intervention period)
Population: All randomized women except one woman in the Gynophilus LP group who withdrew immediately after enrollment.
Measure: Number (95% Confidence Interval); unit: Incidence: events per PY at risk
Groups:
- Control Arm: Behavioral counseling only
- Metronidazole Arm: Counseling plus 2-month intermittent use of oral metronidazole
- Ecologic Femi+ Arm: Counseling plus 2-month intermittent use of Ecologic Femi+ vaginal probiotic capsule
- Gynophilus LP Arm: Counseling plus 2-month intermittent use of Gynophilus LP vaginal probiotic tablet
Arm/Group | Control Arm | Metronidazole Arm | Ecologic Femi+ Arm | Gynophilus LP Arm
Number analyzed (Participants) | 17 | 17 | 17 | 16
Incidence: events per PY at risk | 1.10 [0.35 to 3.41] | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0]

4. Primary Outcome: Vaginal Candidiasis Incidence by Wet Mount Microscopy
Description: A wet mount is a smear of vaginal fluid on a microscopy slide, which is examined under a microscope. Yeasts are visible without staining. The definition of vaginal candidiasis was any yeast visible on the wet mount. Symptomatic vaginal candidiasis was considered a safety outcome because treatment of bacterial vaginosis often results in vaginal candidiasis. Intent-to-treat (ITT) analysis with person-years (PY) at risk as the denominator of all incidence rates.
Time Frame: 6 months: 2 months intervention period plus 4 months after intervention cessation
Population: All randomized women except one woman in the Gynophilus LP group who withdrew immediately after enrollment.
Measure: Number (95% Confidence Interval); unit: Incidence: events per PY at risk
Arm/Group | Control | Oral Metronidazole | Ecologic Femi+ | Gynophilus LP
Number analyzed (Participants) | 17 | 17 | 17 | 16
Incidence: events per PY at risk | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0]

5. Secondary Outcome: Vaginal Microbiota Composition by Illumina HiSeq Sequencing: Lactobacillus Genus Concentration
Description: The vaginal microbiota sequencing results are exploratory and full data can be found in a manuscript on the BioRxiv preprint server. The most important outcome is the concentration of Lactobacillus genus in vaginal samples taken at the end of the intervention period (M2 visit).
Time Frame: 2 months (intervention period)
Population: All randomized women except for one woman in Gynophilus LP who withdrew immediately after enrollment, using lactobacillus concentration in log10 copies per microliter at the M2 visit (at the time of intervention cessation).
Measure: Mean (95% Confidence Interval); unit: Lactobacillus log10 copies/microliter
Arm/Group | Control | Oral Metronidazole | Ecologic Femi+ | Gynophilus LP
Number analyzed (Participants) | 17 | 17 | 17 | 16
Lactobacillus log10 copies/microliter | 3.86 [2.53 to 5.19] | 5.21 [4.27 to 6.14] | 5.30 [4.97 to 5.63] | 4.68 [3.55 to 5.81]

6. Other Pre Specified Outcome: Feasibility/Acceptability of Vaginal Probiotic Use by Structured Face-to-face Interview
Description: Full results have been submitted for publication. Adherence was measured at D7, M1, and M2 visits, and a summary measure over the entire period was calculated (available for women using oral metronidazole, Ecologic Femi+, or Gynophilus LP). After the 2-month intervention period, women using vaginal probiotics (Ecologic Femi+ or Gynophilus LP) were asked structured questions about their experiences with product use.
Time Frame: 2 months (intervention period)
Population: Adherence data are available for all randomized women except one woman in the Gynophilus LP group who withdrew immediately after enrollment. Acceptability data are available for all women randomized to the two vaginal probiotics groups except two women in the Gynophilus LP group (another woman withdrew prior to the Month 2 visit).
Measure: Count of Participants; unit: Participants
Arm/Group | Oral Metronidazole | Ecologic Femi+ | Gynophilus LP
Number analyzed (Participants) | 17 | 17 | 16
Participants
  Perfect (100%) overall adherence | 12 | 10 | 8
  Overall adherence ≥90% | 14 | 15 | 11
  Overall adherence ≥80% | 15 | 17 | 13
  Probiotic insertion as "very comfortable": number analyzed (Participants) | 0 | 17 | 15
  Probiotic insertion as "very comfortable" |  | 17 | 15
  Probiotic insertion became easier over time: number analyzed (Participants) | 0 | 17 | 15
  Probiotic insertion became easier over time |  | 17 | 15

ADVERSE EVENTS:
Time Frame: 6 months: during the 2-month intervention period and up to 4 months after intervention cessation
Description: The definition of adverse events does not differ from the clinicaltrials.gov definitions.
Arm/Group | Control | Oral Metronidazole | Ecologic Femi+ | Gynophilus LP
All-Cause Mortality (participants affected / at risk) | 0/17 | 0/17 | 0/17 | 0/17
Serious Adverse Events (participants affected / at risk) | 0/17 | 1/17 | 1/17 | 0/17
Other Adverse Events (participants affected / at risk) | 2/17 | 2/17 | 2/17 | 3/17
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Control (N=17) | Oral Metronidazole (N=17) | Ecologic Femi+ (N=17) | Gynophilus LP (N=17)
Typhoid fever (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — A participant was hospitalized with typhoid fever during the study; this occurred after the intervention period.
Malaria during pregnancy (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — A participant was hospitalized with malaria (while pregnant) during the study; this occurred after the intervention period.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Control (N=17) | Oral Metronidazole (N=17) | Ecologic Femi+ (N=17) | Gynophilus LP (N=17)
Burning when passing urine (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Genital burning (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Genital itching (Reproductive system and breast disorders) | 2 (2) | 2 (2) | 2 (2) | 2 (2)
Pain during sex (Reproductive system and breast disorders) | 1 (1) | 2 (2) | 0 (0) | 1 (1)
Lower abdominal pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Unusual vaginal discharge (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sores in the genital and/or anal area (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
The two most important limitations were the modest sample size (this trial was funded as a pilot trial) and our inability to exclude women with gonorrhea and/or chlamydia infection at the time of randomization (due to slow testing turn-around).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2015-04-22): https://cdn.clinicaltrials.gov/large-docs/65/NCT02459665/Prot_000.pdf
  • Statistical Analysis Plan (2016-09-16): https://cdn.clinicaltrials.gov/large-docs/65/NCT02459665/SAP_001.pdf